CLINICAL TRIAL: NCT02794701
Title: Comprehensive Risk Assessment of People With Silicosis: A Population-based Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Yu CHENG, post-doctoral fellow, Chinese University of Hong Kong
Other Study IDs: CRE-2015.499
Record Dates: First submitted 2016-05-30; First posted 2016-06-09 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Silicosis
MeSH Terms: conditions — Silicosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- people with silicosis
  Interventions: Other: People with silicosis

INTERVENTIONS:
Other: People with silicosis

SUMMARY:
Objectives: This study aims to explore the risk profiles among people with silicosis in Hong Kong underpinned by the Pittsburgh Mind-Body Center model.

Design and subjects: This study will adopt a cross-sectional study design with sampling stratified by participants' degree of incapability. 320 Chinese people diagnosed with silicosis and registered with the Pneumoconiosis Compensation Fund Board will be recruited.

Data collection: A demographic data sheet and the St. George's Respiratory Questionnaire will be used to collect the socio-demographic and clinical characteristics of the participants. The behavioral factors (smoking, drinking, physical activity level, consumption of vegetable and fruits and plasma vitamin C level) as well as the psychological risk factors (anxiety and depressive symptoms, and social support) will be examined by validated questionnaires. Biological and physiological parameters, including insulin resistance, C-reactive protein, hemoglobin, fasting blood glucose and lipid profiles, will be ascertained by fasting blood sample.

Data analysis and expected outcomes: The findings of this study will create the database profile of the physical, psychosocial and disease specific aspects among people with silicosis in Hong Kong, subsequently forming the empirical basis of an intervention to tackle the identified modifiable risks among them.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese-speaking residents and Chinese ethnicity;
* diagnosis of silicosis and confirmed by the Pneumoconiosis Medical Board
* registered with the Pneumoconiosis Compensation Fund Board (PCFB); and
* able and willing to give informed written consent

Exclusion Criteria:

* With medically diagnosed mental illness, including major depression, or
* with active pulmonary tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 390 eligible participants registered with the Pneumoconiosis Compensation Fund Board will be recruited with stratification by their degree of incapacity [(i) <30%, (ii) 30% - 60%, and (iii) >60%], in which the minimal number of participants in each strata will be 30.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Respiratory symptoms and related physical limitation | baseline
  examined by Hong Kong Chinese version of St. George's Respiratory Questionnaire
Psychological status | baseline
  Anxiety and depression symptoms measured by the Chinese version of Hospital Anxiety and Depression Scale
Quality of life | baseline
  examined by the SF-12v2
Social support | baseline
  measured by the Chinese version of six-item Social Support Questionnaire
Body mass index | baseline
  BMI in kg/m^2
waist circumference | baseline
  WC in cm
12-hour fasting lipid profile | baseline
  total-cholesterol, HDL-Cholesterol, LDL-cholesterol and triglycerides (in mmol/L)
12-hour fasting glucose | baseline
  FG in mmol/L
fasting insulin level | baseline
  insulin in pmol/L
12 hour fasting ascorbic acid level | baseline
  vit-C in mg/dL
fasting high sensitivity C-reactive protein level | baseline
  hs-CRP in mg/L
hemoglobin level | baseline
  hemoglobin in g/dL
smoking and drinking habits, vegetable and fruit intake | baseline
  questions adopted from the Behavioral Risk Factor Surveillance of the Department of Health, Hong Kong SAR
Physical activity level | baseline
  measured by the International Physical Activity Questionnaire - Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yu CHENG, PhD, RN, Principal Investigator — The Nethersole School of Nursing, Chinese University of Hong Kong
Locations (1):
- The Nethersole School of Nursing, Chinese University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No